CLINICAL TRIAL: NCT03471871
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Evaluate the Respiratory Safety of Lemborexant in Adult and Elderly Healthy Subjects and Adult and Elderly Subjects With Mild Obstructive Sleep Apnea
Brief Title: Study to Evaluate the Respiratory Safety of Lemborexant in Adult and Elderly Healthy Subjects and Adult and Elderly Subjects With Mild Obstructive Sleep Apnea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: E2006-A001-102
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2018-07

CONDITIONS: Obstructive Sleep Apnea; Healthy Subjects
Keywords: Elderly Healthy Subjects; Adult Healthy Subjects; Lemborexant; Respiratory Safety; Peripheral Oxygen Saturation; Total Sleep Time
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — lemborexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- HV Cohort,Sequence A:Placebo,Lemborexant 10mg,Lemborexant 25mg (Experimental): Eligible healthy adult and elderly participants will receive lemborexant-matched placebo (3 matched tablets) on the night of Day 1 of Treatment Period 1, followed by lemborexant 10 mg (1 lemborexant 10 mg tablet and 2 matching placebo tablets) on the night of Day 1 of Treatment Period 2, and then lemborexant 25 mg (2 lemborexant 10 mg tablets and 1 lemborexant 5 mg tablet) on the night of Day 1 of Treatment Period 3. A washout period of 14 days was maintained between each Treatment Period.
  Interventions: Drug: Placebo; Drug: Lemborexant 10 mg; Drug: Lemborexant 25 mg
- HV Cohort,Sequence B:Lemborexant 10mg,Lemborexant 25mg,Placebo (Experimental): Eligible healthy adult and elderly participants will receive lemborexant 10 mg (1 lemborexant 10 mg tablet and 2 matching placebo tablets) on the night of Day 1 of Treatment Period 1, followed by lemborexant 25 mg (2 lemborexant 10 mg tablets and 1 lemborexant 5 mg tablet) on the night of Day 1 of Treatment Period 2, and then lemborexant-matched placebo (3 matched tablets) on the night of Day 1 of Treatment Period 3. A washout period of 14 days was maintained between each Treatment Period.
  Interventions: Drug: Placebo; Drug: Lemborexant 10 mg; Drug: Lemborexant 25 mg
- HV Cohort,Sequence C:Lemborexant 25mg,Placebo,Lemborexant 10mg (Experimental): Eligible healthy adult and elderly participants will receive lemborexant 25 mg (2 lemborexant 10 mg tablet and 1 lemborexant 5 mg tablet) on the night of Day 1 of Treatment Period 1, followed by lemborexant-matched placebo (3 matched tablets) on the night of Day 1 of Treatment Period 2, and then lemborexant 10 mg (1 lemborexant 10 mg tablet and 2 matching placebo tablets) on the night of Day 1 of Treatment Period 3. A washout period of 14 days was maintained between each Treatment Period.
  Interventions: Drug: Placebo; Drug: Lemborexant 10 mg; Drug: Lemborexant 25 mg
- OSA Cohort, Sequence D: Placebo, Lemborexant 10mg (Experimental): Eligible adult and elderly participants with mild OSA will receive one lemborexant-matched placebo tablet on the night of Day 1 through Day 8 of Treatment Period 1, followed by one lemborexant 10 mg tablet on the night of Day 1 through Day 8 of Treatment Period 2. A washout period of 14 days was maintained between each Treatment Period.
  Interventions: Drug: Placebo; Drug: Lemborexant 10 mg
- OSA Cohort, Sequence E: Lemborexant 10mg, Placebo (Experimental): Eligible adult and elderly participants with mild OSA will receive one lemborexant 10 mg tablet on the night of Day 1 through Day 8 of Treatment Period 1, followed by one lemborexant-matched placebo tablet on the night of Day 1 through Day 8 of Treatment Period 2. A washout period of 14 days was maintained between each Treatment Period.
  Interventions: Drug: Placebo; Drug: Lemborexant 10 mg

INTERVENTIONS:
Drug: Placebo — HV: Lemborexant-matched oral placebo will be administered at bedtime in the clinic (within 5 minutes of lights off).
  Arms: HV Cohort,Sequence A:Placebo,Lemborexant 10mg,Lemborexant 25mg; HV Cohort,Sequence B:Lemborexant 10mg,Lemborexant 25mg,Placebo; HV Cohort,Sequence C:Lemborexant 25mg,Placebo,Lemborexant 10mg
Drug: Lemborexant 10 mg — HV: 10 mg oral lemborexant will be administered at bedtime in the clinic (within 5 minutes of lights off).
  Arms: HV Cohort,Sequence A:Placebo,Lemborexant 10mg,Lemborexant 25mg; HV Cohort,Sequence B:Lemborexant 10mg,Lemborexant 25mg,Placebo; HV Cohort,Sequence C:Lemborexant 25mg,Placebo,Lemborexant 10mg
Drug: Lemborexant 25 mg — HV: 25 mg oral lemborexant will be administered at bedtime in the clinic (within 5 minutes of lights off).
  Arms: HV Cohort,Sequence A:Placebo,Lemborexant 10mg,Lemborexant 25mg; HV Cohort,Sequence B:Lemborexant 10mg,Lemborexant 25mg,Placebo; HV Cohort,Sequence C:Lemborexant 25mg,Placebo,Lemborexant 10mg
Drug: Placebo — OSA: Lemborexant-matched oral placebo will be administered at bedtime in the clinic (within 5 minutes of lights off) in the evening of Days 1 and 8. On Days 2 to 7, participants will take study drug at home, immediately (within 5 minutes) of the time they intend to try to sleep.
  Arms: OSA Cohort, Sequence D: Placebo, Lemborexant 10mg; OSA Cohort, Sequence E: Lemborexant 10mg, Placebo
Drug: Lemborexant 10 mg — OSA: 10 mg oral lemborexant will be administered at bedtime in the clinic (within 5 minutes of lights off) in the evening of Days 1 and 8. On Days 2 to 7, participants will take study drug at home, immediately (within 5 minutes) of the time they intend to try to sleep.
  Arms: OSA Cohort, Sequence D: Placebo, Lemborexant 10mg; OSA Cohort, Sequence E: Lemborexant 10mg, Placebo

SUMMARY:
This study will be conducted to determine whether lemborexant as compared to placebo decreases the peripheral oxygen saturation during total sleep time in healthy adult and elderly participants after a single dose of treatment and to determine whether it increases the apnea-hypopnea index after single and multiple doses of treatment in adult and elderly participants with mild obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
Healthy Volunteer (HV) Cohort:

The HV Cohort comprises a randomized, double-blind, placebo-controlled, 3-period crossover study. Eligible healthy adult and elderly participants will be randomized to treatment sequence A, B, or C, each consisting of 3 Treatment Periods, each of one night's duration, in which participants will receive a single dose of lemborexant 10 milligrams (mg), or lemborexant 25 mg, or placebo. Treatment Periods will be separated by a washout interval of at least 14 days. A sufficient number of participants will be randomized to ensure that 8 evaluable adult participants (<65 years) and 4 evaluable elderly participants (≥65 years) complete the study.

OSA Cohort:

The OSA Cohort comprises a multiple-dose, randomized, double-blind, placebo-controlled, 2-period crossover study. Adult and elderly participants with mild OSA will be randomized to treatment sequence D or E, each consisting of 2 Treatment Periods, each of 8 nights' duration, in which participants will receive lemborexant 10 mg or placebo. The Treatment Periods will be separated by a washout interval of at least 14 days. A sufficient number of participants will be randomized to ensure that 20 evaluable adult participants (<65 years) and 10 evaluable elderly participants (≥65 years) complete the study.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in this study:

* Male or female, age ≥18 years and ≤90 years at the time of informed consent
* Voluntary agreement and ability to provide written informed consent
* Reports habitually sleeping for at least 5.5 hours per night
* Agrees to stay in bed for 7 hours per night for the duration of treatment
* Reports habitual bedtime between 21:00 and 01:00
* Peripheral capillary oxygen saturation (SpO2) ≥94% assessed as part of vital signs at Screening Visit 1

Additional Inclusion Criteria (Healthy Volunteer [HV] Cohort):

* Body mass index (BMI) less than or equal to 32 kilograms per meters squared (kg/m^2)
* On screening polysomnography (PSG) (Screening Visit 2): apnea-hypopnea index (AHI) <5

Additional Inclusion Criteria (Obstructive Sleep Apnea [OSA] Cohort):

* BMI ≤40 kg/m^2
* OSA, diagnosed according to the criteria of the International Classification of Sleep Disorders, version 3
* On Screening PSG: AHI ≥5 to <15 (mild severity)

Exclusion Criteria:

* A current diagnosis of restless legs syndrome, periodic limb movement disorder, circadian rhythm sleep disorder, or narcolepsy
* Reports symptoms potentially related to narcolepsy, that in the clinical opinion of the investigator indicate the need for referral for a diagnostic evaluation for the presence of narcolepsy
* A history of a parasomnia or parasomnia observed on the Screening PSG that in the investigator's opinion makes the participant unsuitable for the study
* Periodic Limb Movement with Arousal Index (PLMAI) as measured on the Screening PSG:

  1. Age 18 to <65 years: PLMAI ≥10
  2. Age ≥65 years: PLMAI >15
* History of or suspected drug or alcohol use disorder within approximately 2 previous years
* A positive urine drug test or breath alcohol test at Screening or Baseline, or unwilling to refrain from use of recreational drugs during the study
* Known to be human immunodeficiency virus positive
* Active viral hepatitis (B or C) as demonstrated by positive viral serology at Screening
* A prolonged QT/corrected QT (QTc) interval (QT interval corrected for heart rate using Fridericia's formula [QTcF] >450 milliseconds [ms]) as demonstrated by a repeated electrocardiogram (ECG) at Screening (repeated if initial ECG indicates a QTcF interval >450 ms)
* Comorbid nocturia resulting in the need to get out of bed to use the bathroom more than 3 times during the night
* Any history of medical or psychiatric condition that in the opinion of the investigator could affect the participant's safety or interfere with the study assessments
* Any suicidal ideation with intent to act with or without a plan, current or within 6 months before the Columbia - Suicide Severity Rating Scale (C-SSRS) administration during the Screening (e.g., answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the C-SSRS
* Any suicidal behavior (per the Suicidal Behavior section of the C-SSRS) within 10 years of Screening
* Scheduled for surgery during the study that requires general anesthesia or administration of prohibited medications
* Used any prohibited prescription or over-the-counter medications within 1 week or 5 half-lives, whichever is longer, before the Screening PSG
* Hypersensitivity to lemborexant or excipients
* Currently enrolled in another interventional clinical trial or used any investigational drug or device within 30 days or 5 times the half-life, whichever is longer preceding informed consent
* Previously participated in other clinical trial of lemborexant
* Is unable to avoid working a night shift within 2 weeks before the Screening PSG, or between the Screening PSG and End-of-Study
* Has travelled across 3 or more time zones in the week prior to Screening, or plans to travel across more than 3 time zones during the study
* Clinically significant findings based on vital signs, physical examination, ECG, or clinical laboratory tests

Additional Exclusion Criteria (HV Cohort):

* Any valid event of SpO2 <90% during the Screening PSG
* Current evidence of a clinically significant, active respiratory disorder. This includes bronchiectasis, emphysema, asthma, chronic obstructive pulmonary disease, or any other pulmonary disorder identified by review of medical history, physical examination, and which in the opinion of the investigator, could compromise the participant's safety or interfere with study assessments
* Presence of significant illness (including insomnia) that requires treatment or may influence the study assessments (e.g., psychiatric disorders, disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, cardiovascular system, or a congenital abnormality), malignancy within the past 5 years (other than adequately treated basal cell carcinoma or in situ carcinoma of the cervix), or chronic pain that in the opinion of the investigator could interfere with the study assessments. Participants for whom a sedating drug would be contraindicated for safety reasons because of the participant's occupation or activities are also excluded

Additional Exclusion Criteria (OSA Cohort):

* SpO2 less than 80% for ≥ 5% of total sleep time during the Screening PSG
* Uses or plans to use of continuous positive airway pressure device or dental appliance within 2 weeks of the Screening PSG (Screening Visit 2) or during the study
* Current evidence of a clinically significant, active respiratory disorder other than OSA. This includes bronchiectasis, emphysema, asthma, chronic obstructive pulmonary disease or any other pulmonary disorder identified by review of medical history, physical examination, and which in the opinion of the investigator, could compromise the participant's safety or interfere with study assessments
* Current evidence of other clinically significant disease (e.g., psychiatric disorders, disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, cardiovascular system, or a congenital abnormality), malignancy within the past 5 years (other than adequately treated basal cell carcinoma or in situ carcinoma of the cervix), or chronic pain that in the opinion of the investigator could affect the participant's safety or interfere with the study assessments. Participants for whom a sedating drug would be contraindicated for safety reasons because of the participant's occupation or activities are also excluded. Participants with insomnia disorder, who complain of difficulties with sleep onset and/or sleep maintenance, are eligible provided that they meet this criterion. Note that medications to treat insomnia are prohibited.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - PACT, Glendale, Arizona
  - Pulmonary Associates, PA, Phoenix, Arizona
  - Pacific Research Network. LLC, San Diego, California
  - PAB Clinical Research, Brandon, Florida
  - Research Centers of America, Hollywood, Florida
  - Neurotrials Research, Inc, Atlanta, Georgia
  - The Center for Sleep & Wake Disorders, Chevy Chase, Maryland
  - Advarra, Columbia, Maryland
  - Clinilabs Drug Development, New York, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio

REFERENCES:
- [Derived] Khullar A, Boulos MI, Mak MSB, Moline M, Cheng JY, Hall N. Effect of lemborexant on sleep parameters and architecture in adult and elderly participants with mild-to-severe obstructive sleep apnea. Sleep Med. 2025 Oct;134:106757. doi: 10.1016/j.sleep.2025.106757. Epub 2025 Aug 18. PMID 40848323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in the United States from February 21, 2018 to August 3, 2018.
Pre-assignment Details: In healthy volunteer (HV) cohort, 39 participants were screened and enrolled, of which 22 were screen failures, 17 were randomized to receive treatment. In obstructive sleep apnea (OSA) cohort, 107 participants were screened and enrolled, of which 68 were screen failures, 39 were randomized to receive treatment. Total participants enrolled=146
Groups:
- HV Cohort,Sequence A:Placebo,Lemborexant 10mg,Lemborexant 25mg: Eligible healthy adult and elderly participants received lemborexant-matched placebo (3 placebo tablets), orally, once, in the evening (within 5 minutes of lights off) of Day 1 of Treatment Period 1, followed by lemborexant 10 mg (milligram) (1 lemborexant 10 mg tablet and 2 matching placebo tablets [to maintain blind]), orally, once, in the evening (within 5 minutes of lights off) of Day 1 of Treatment Period 2, and then lemborexant 25 mg (2 lemborexant 10 mg tablets and 1 lemborexant 5 mg tablet), orally, once, in the evening (within 5 minutes of lights off) of Day 1 of Treatment Period 3. A washout period of 14 days was maintained between each treatment period.
- HV Cohort,Sequence B:Lemborexant 10mg,Lemborexant 25mg,Placebo: Eligible healthy adult and elderly participants received lemborexant 10 mg (1 lemborexant 10 mg tablet and 2 matching placebo tablets [to maintain blind]), orally, once, in the evening (within 5 minutes of lights off) of Day 1 of Treatment Period 1, followed by lemborexant 25 mg (2 lemborexant 10 mg tablets and 1 lemborexant 5 mg tablet), orally, once, in the evening (within 5 minutes of lights off) of Day 1 of Treatment Period 2, and then lemborexant-matched placebo (3 placebo tablets), orally, once, in the evening (within 5 minutes of lights off) of Day 1 of Treatment Period 3. A washout period of 14 days was maintained between each treatment period.
- HV Cohort,Sequence C:Lemborexant 25mg,Placebo,Lemborexant 10mg: Eligible healthy adult and elderly participants received lemborexant 25 mg (2 lemborexant 10 mg tablets and 1 lemborexant 5 mg tablet), orally, once, in the evening (within 5 minutes of lights off) of Day 1 of Treatment Period 1, followed by lemborexant-matched placebo (3 placebo tablets), orally, once, in the evening (within 5 minutes of lights off) of Day 1 of Treatment Period 2, and then lemborexant 10 mg (1 lemborexant 10 mg tablet and 2 matching placebo tablets [to maintain blind]), orally, once, in the evening (within 5 minutes of lights off) of Day 1 of Treatment Period 3. A washout period of 14 days was maintained between each treatment period.
- OSA Cohort, Sequence D: Placebo, Lemborexant 10mg: Eligible adult and elderly participants with mild OSA received one lemborexant-matched placebo, tablet, orally, once, in the evening (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Period 1, followed by one lemborexant 10 mg, tablet, orally, once, in the evening (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Period 2. A washout period of 14 days was maintained between each treatment period.
- OSA Cohort, Sequence E: Lemborexant 10mg, Placebo: Eligible adult and elderly participants with mild OSA received one lemborexant 10 mg, tablet, orally, once in the evening of Day 1 through Day 8 of Treatment Period 1, followed by one lemborexant-matched placebo, tablet, orally, once, in the evening of Day 1 through Day 8 of Treatment Period 2. A washout period of 14 days was maintained between each treatment period.
Period: Treatment Period 1(HV:1 Day, OSA:8 Days)
Arm/Group | HV Cohort,Sequence A:Placebo,Lemborexant 10mg,Lemborexant 25mg | HV Cohort,Sequence B:Lemborexant 10mg,Lemborexant 25mg,Placebo | HV Cohort,Sequence C:Lemborexant 25mg,Placebo,Lemborexant 10mg | OSA Cohort, Sequence D: Placebo, Lemborexant 10mg | OSA Cohort, Sequence E: Lemborexant 10mg, Placebo
Started | 6 | 5 | 6 | 19 | 20
Treated | 6 | 5 | 6 | 18 | 20
Completed | 6 | 5 | 5 | 18 | 19
Not Completed | 0 | 0 | 1 | 1 | 1
Not completed — Work Demand: Return to work | 0 | 0 | 1 | 0 | 0
Not completed — Protocol deviation | 0 | 0 | 0 | 1 | 1
Period: Washout Period 1 (14 Days)
Arm/Group | HV Cohort,Sequence A:Placebo,Lemborexant 10mg,Lemborexant 25mg | HV Cohort,Sequence B:Lemborexant 10mg,Lemborexant 25mg,Placebo | HV Cohort,Sequence C:Lemborexant 25mg,Placebo,Lemborexant 10mg | OSA Cohort, Sequence D: Placebo, Lemborexant 10mg | OSA Cohort, Sequence E: Lemborexant 10mg, Placebo
Started | 6 | 5 | 5 | 18 | 19
Completed | 6 | 5 | 5 | 18 | 19
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2(HV:1 Day, OSA:8 Days)
Arm/Group | HV Cohort,Sequence A:Placebo,Lemborexant 10mg,Lemborexant 25mg | HV Cohort,Sequence B:Lemborexant 10mg,Lemborexant 25mg,Placebo | HV Cohort,Sequence C:Lemborexant 25mg,Placebo,Lemborexant 10mg | OSA Cohort, Sequence D: Placebo, Lemborexant 10mg | OSA Cohort, Sequence E: Lemborexant 10mg, Placebo
Started | 6 | 5 | 5 | 18 | 19
Completed | 6 | 5 | 5 | 18 | 18
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 1
Period: Washout Period 2 (14 Days)
Arm/Group | HV Cohort,Sequence A:Placebo,Lemborexant 10mg,Lemborexant 25mg | HV Cohort,Sequence B:Lemborexant 10mg,Lemborexant 25mg,Placebo | HV Cohort,Sequence C:Lemborexant 25mg,Placebo,Lemborexant 10mg | OSA Cohort, Sequence D: Placebo, Lemborexant 10mg | OSA Cohort, Sequence E: Lemborexant 10mg, Placebo
Started | 6 | 5 | 5 | 0 (0=not applicable, as OSA cohort was treated till Treatment Period 2, then directly followed up.) | 0 (0=not applicable, as OSA cohort was treated till Treatment Period 2, then directly followed up.)
Completed | 6 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3: ( HV:1 Day)
Arm/Group | HV Cohort,Sequence A:Placebo,Lemborexant 10mg,Lemborexant 25mg | HV Cohort,Sequence B:Lemborexant 10mg,Lemborexant 25mg,Placebo | HV Cohort,Sequence C:Lemborexant 25mg,Placebo,Lemborexant 10mg | OSA Cohort, Sequence D: Placebo, Lemborexant 10mg | OSA Cohort, Sequence E: Lemborexant 10mg, Placebo
Started | 6 | 5 | 5 | 0 | 0
Completed | 6 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Follow Up (14 Days for Both HV and OSA)
Arm/Group | HV Cohort,Sequence A:Placebo,Lemborexant 10mg,Lemborexant 25mg | HV Cohort,Sequence B:Lemborexant 10mg,Lemborexant 25mg,Placebo | HV Cohort,Sequence C:Lemborexant 25mg,Placebo,Lemborexant 10mg | OSA Cohort, Sequence D: Placebo, Lemborexant 10mg | OSA Cohort, Sequence E: Lemborexant 10mg, Placebo
Started | 6 | 5 | 5 | 18 (OSA cohort was treated till Treatment Period 2 only and then entered in follow up period.) | 18 (OSA cohort was treated till Treatment Period 2 only and then entered in follow up period.)
Completed | 6 | 5 | 5 | 17 | 17
Not Completed | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 1
Not completed — Did Return to Clinic | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data has been presented as per study cohorts (HV and OSA) involved in the study.
Groups:
- HV Cohort: Eligible healthy adult and elderly participants received lemborexant-matched placebo (3 placebo tablets), lemborexant 10 mg (1 lemborexant 10 mg tablet and 2 matching placebo tablets [to maintain blind]) or lemborexant 25 mg (2 lemborexant 10 mg tablets and 1 lemborexant 5 mg tablet), orally, once, in the evening (within 5 minutes of lights off) of Day 1 in the respective Treatment Period 1, 2 or 3. A washout period of 14 days was maintained between each treatment period.
- OSA Cohort: Eligible adult and elderly participants with mild OSA received one lemborexant-matched placebo or one lemborexant 10 mg, tablets, orally, once, in the evening (within 5 minutes of lights off) of Day 1 through Day 8 in the respective Treatment Period 1 or 2. A washout period of 14 days was maintained between each treatment period.
- Total: Total of all reporting groups
Arm/Group | HV Cohort | OSA Cohort | Total
Number analyzed (Participants) | 17 | 39 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 26 | 36
  >=65 years | 7 | 13 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 24 | 36
  Male | 5 | 15 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 16 | 17
  Not Hispanic or Latino | 16 | 23 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 3 | 11
  White | 9 | 35 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: HV Cohort: Peripheral Oxygen Saturation (SpO2) During Total Sleep Time (TST) on Day 1 of Treatment
Description: SpO2 is an estimate of the amount of oxygen in the blood. It is the percentage of hemoglobin containing oxygen compared to the total amount of hemoglobin in the blood (that is, oxygenated hemoglobin versus oxygenated and non-oxygenated hemoglobin). SpO2 was monitored by noninvasive method known as transmissive pulse oximetry. TST was defined as the total time asleep in minutes using polysomnography (PSG).
Time Frame: Day 1
Population: Pharmacodynamic (PD) analysis set included group of participants who received at least 1 dose of study drug in each treatment periods and who had sufficient PD data to derive at least 1 primary PD parameter.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Groups:
- HV Cohort: Placebo: Eligible healthy adult and elderly participants received lemborexant-matched placebo (3 placebo tablets), orally, once, in the evening (within 5 minutes of lights off) of Day 1 in the respective Treatment Period 1, 2 or 3.
- HV Cohort: Lemborexant 10 mg: Eligible healthy adult and elderly participants received lemborexant 10 mg (1 lemborexant 10 mg tablet and 2 matching placebo tablets [to maintain blind]), orally, once, in the evening (within 5 minutes of lights off) of Day 1 in the respective Treatment Period 1, 2 or 3.
- HV Cohort: Lemborexant 25 mg: Eligible healthy adult and elderly participants received lemborexant 25 mg (2 lemborexant 10 mg tablets and 1 lemborexant 5 mg tablet), orally, once, in the evening (within 5 minutes of lights off) of Day 1 in the respective Treatment Period 1, 2 or 3.
Arm/Group | HV Cohort: Placebo | HV Cohort: Lemborexant 10 mg | HV Cohort: Lemborexant 25 mg
Number analyzed (Participants) | 16 | 16 | 16
percentage of oxygen saturation | 95.34 (0.900) | 95.00 (1.283) | 95.07 (1.311)
Statistical Analysis 1: Comparison: HV Cohort: Placebo vs HV Cohort: Lemborexant 10 mg; Test type: Other; p = 0.099, Mixed effect model — P-Value was at the 0.05 level of significance; SPO2 was analyzed by mixed effect model, which included fixed effects for sequence, period, treatment a random effect for participant within sequence; Least squares (LS) mean difference = -0.36, 95% CI 2-sided [-0.78 to 0.07]
Statistical Analysis 2: Comparison: HV Cohort: Placebo vs HV Cohort: Lemborexant 25 mg; Test type: Other; p = 0.176, Mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.29, 95% CI 2-sided [-0.72 to 0.14]

2. Primary Outcome: OSA Cohort: Apnea-Hypopnea Index (AHI) on Day 8 of Treatment
Description: The AHI is the number of apneas and hypopneas per hour of sleep. AHI less than 5 is considered normal. An AHI from 5 to 14 denotes mild sleep apnea, 15 to 30 is moderate, while a greater than 30 AHI is considered severe.
Time Frame: Day 8
Population: PD analysis set included group of participants who received at least 1 dose of study drug in each treatment periods and who had sufficient PD data to derive at least 1 primary PD parameter. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: events (apnea plus hyponea) per hour
Groups:
- OSA Cohort: Placebo: Eligible adult and elderly participants with mild OSA received one lemborexant-matched placebo, tablet, orally, once, in the evening (within 5 minutes of lights off) of Day 1 through Day 8 in the respective Treatment Period 1 or 2.
- OSA Cohort: Lemborexant 10 mg: Eligible adult and elderly participants with mild OSA received one lemborexant 10 mg, tablet, orally, once, in the evening (within 5 minutes of lights off) of Day 1 through Day 8 in the respective Treatment Period 1 or 2.
Arm/Group | OSA Cohort: Placebo | OSA Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 35 | 37
events (apnea plus hyponea) per hour | 10.03 (6.799) | 9.99 (5.878)
Statistical Analysis 1: Comparison: OSA Cohort: Placebo vs OSA Cohort: Lemborexant 10 mg; Test type: Other; p = 0.948, Mixed effect model — P-Value was at the 0.05 level of significance; AHI was analyzed by mixed effect model, which included fixed effects for sequence, period, treatment a random effect for participant within sequence; LS mean difference = -0.06, 95% CI 2-sided [-1.95 to 1.83]

3. Secondary Outcome: HV Cohort: AHI on Day 1 of Treatment
Description: as for outcome 2
Time Frame: Day 1
Population: PD analysis set included group of participants who received at least 1 dose of study drug in each treatment periods and who had sufficient PD data to derive at least 1 primary PD parameter.
Measure: Mean (Standard Deviation); unit: events (apnea plus hyponea) per hour
Arm/Group | HV Cohort: Placebo | HV Cohort: Lemborexant 10 mg | HV Cohort: Lemborexant 25 mg
Number analyzed (Participants) | 16 | 16 | 16
events (apnea plus hyponea) per hour | 4.69 (8.183) | 5.29 (10.484) | 3.55 (6.585)
Statistical Analysis 1: Comparison: HV Cohort: Placebo vs HV Cohort: Lemborexant 10 mg; Test type: Other; p = 0.639, Mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 2, analysis 1]; LS mean difference = 0.52, 95% CI 2-sided [-1.72 to 2.76]
Statistical Analysis 2: Comparison: HV Cohort: Placebo vs HV Cohort: Lemborexant 25 mg; Test type: Other; p = 0.297, mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 2, analysis 1]; LS mean difference = -1.16, 95% CI 2-sided [-3.40 to 1.08]

4. Secondary Outcome: OSA Cohort: AHI on Day 1 of Treatment
Description: as for outcome 2
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: events (apnea plus hyponea) per hour
Arm/Group | OSA Cohort: Placebo | OSA Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 37 | 36
events (apnea plus hyponea) per hour | 10.24 (7.094) | 10.29 (6.681)
Statistical Analysis 1: Comparison: OSA Cohort: Placebo vs OSA Cohort: Lemborexant 10 mg; Test type: Other; p = 0.979, Mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 2, analysis 1]; LS mean difference = -0.03, 95% CI 2-sided [-2.22 to 2.17]

5. Secondary Outcome: HV Cohort: Percentage of TST During Which SpO2 Was Less Than (<) 90 Percent (%), 85 % and 80 % on Day 1 of Treatment
Description: TST was defined as the total time asleep in minutes using PSG. SpO2 is an estimate of the amount of oxygen in the blood. It is the percentage of hemoglobin containing oxygen compared to the total amount of hemoglobin in the blood (that is, oxygenated hemoglobin versus oxygenated and non-oxygenated hemoglobin). SpO2 was monitored by noninvasive method known as transmissive pulse oximetry.
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of TST
Arm/Group | HV Cohort: Placebo | HV Cohort: Lemborexant 10 mg | HV Cohort: Lemborexant 25 mg
Number analyzed (Participants) | 16 | 16 | 16
percentage of TST
  SpO2 <90% | 0.037 (0.0968) | 0.224 (0.3755) | 0.287 (0.5555)
  SpO2 <85% | 0 (0) | 0.004 (0.0109) | 0.047 (0.1516)
  SpO2 <80% | 0 (0) | 0.001 (0.0034) | 0.003 (0.0077)
Statistical Analysis 1: Comparison: HV Cohort: Placebo vs HV Cohort: Lemborexant 10 mg; SpO2 is <90%; Test type: Other; p = 0.095, Mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.185, 95% CI 2-sided [-0.034 to 0.405]
Statistical Analysis 2: Comparison: HV Cohort: Placebo vs HV Cohort: Lemborexant 25 mg; When SpO2 is <90%; Test type: Other; p = 0.030, Mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.245, 95% CI 2-sided [0.025 to 0.464]
Statistical Analysis 3: Comparison: HV Cohort: Placebo vs HV Cohort: Lemborexant 10 mg; SpO2 is <85%; Test type: Other; p = 0.885, Mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.004, 95% CI 2-sided [-0.058 to 0.067]
Statistical Analysis 4: Comparison: HV Cohort: Placebo vs HV Cohort: Lemborexant 25 mg; SpO2 is <85%; Test type: Other; p = 0.158, Mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.044, 95% CI 2-sided [-0.018 to 0.107]
Statistical Analysis 5: Comparison: HV Cohort: Placebo vs HV Cohort: Lemborexant 10 mg; SpO2 is <80%; Test type: Other; p = 0.462, Mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.001, 95% CI 2-sided [-0.002 to 0.005]
Statistical Analysis 6: Comparison: HV Cohort: Placebo vs HV Cohort: Lemborexant 25 mg; SpO2 is <80%; Test type: Other; p = 0.166, Mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.002, 95% CI 2-sided [-0.001 to 0.006]

6. Secondary Outcome: HV Cohort: Percentage of Participants With at Least One Incident of SpO2 <90% for at Least 30 Seconds During TST on Day 1 of Treatment
Description: SpO2 is an estimate of the amount of oxygen in the blood. It is the percentage of hemoglobin containing oxygen compared to the total amount of hemoglobin in the blood (that is, oxygenated hemoglobin versus oxygenated and non-oxygenated hemoglobin). SpO2 was monitored by noninvasive method known as transmissive pulse oximetry. TST was defined as the total time asleep in minutes using PSG.
Time Frame: Day 1
Population: as for outcome 3
Measure: Number; unit: percentage of participant
Arm/Group | HV Cohort: Placebo | HV Cohort: Lemborexant 10 mg | HV Cohort: Lemborexant 25 mg
Number analyzed (Participants) | 16 | 16 | 16
percentage of participant | 31.3 | 31.3 | 37.5

7. Secondary Outcome: OSA Cohort: SpO2 During TST on Day 1 and Day 8 of Treatment
Description: as for outcome 6
Time Frame: Day 1 and Day 8
Population: PD analysis set included group of participants who received at least 1 dose of study drug in each treatment periods and who had sufficient PD data to derive at least 1 primary PD parameter. Here, 'number analyzed' signifies participants who were evaluable for analysis at the specified timepoints.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | OSA Cohort: Placebo | OSA Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 37 | 37
percentage of oxygen saturation
  Day 1: number analyzed (Participants) | 36 | 35
  Day 1 | 94.53 (1.620) | 94.54 (1.470)
  Day 8: number analyzed (Participants) | 35 | 37
  Day 8 | 94.46 (1.316) | 94.65 (1.539)
Statistical Analysis 1: Comparison: OSA Cohort: Placebo vs OSA Cohort: Lemborexant 10 mg; Day 1: Mean SpO2 during TST; Test type: Other; p = 0.699, mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.07, 95% CI 2-sided [-0.31 to 0.46]
Statistical Analysis 2: Comparison: OSA Cohort: Placebo vs OSA Cohort: Lemborexant 10 mg; Day 8: Mean SpO2 during TST; Test type: Other; p = 0.169, mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.25, 95% CI 2-sided [-0.11 to 0.61]

8. Secondary Outcome: OSA Cohort: Percentage of TST During Which the SpO2 is <90%, 85% and 80 % on Day 1 and Day 8 of Treatment
Description: as for outcome 5
Time Frame: Day 1 and Day 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of TST
Arm/Group | OSA Cohort: Placebo | OSA Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 37 | 37
percentage of TST
  Day 1: SpO2 <90%: number analyzed (Participants) | 37 | 36
  Day 1: SpO2 <90% | 1.044 (1.8851) | 1.362 (2.6170)
  Day 1: SpO2 <85%: number analyzed (Participants) | 37 | 36
  Day 1: SpO2 <85% | 0.104 (0.3043) | 0.170 (0.5132)
  Day 1: SpO2 <80%: number analyzed (Participants) | 37 | 36
  Day 1: SpO2 <80% | 0.012 (0.0483) | 0.014 (0.0433)
  Day 8: SpO2 <90%: number analyzed (Participants) | 35 | 37
  Day 8: SpO2 <90% | 1.011 (1.4210) | 1.102 (1.5469)
  Day 8: SpO2 <85%: number analyzed (Participants) | 35 | 37
  Day 8: SpO2 <85% | 0.109 (0.2974) | 0.162 (0.4350)
  Day 8: SpO2 <80%: number analyzed (Participants) | 35 | 37
  Day 8: SpO2 <80% | 0.009 (0.0366) | 0.015 (0.0603)
Statistical Analysis 1: Comparison: OSA Cohort: Placebo vs OSA Cohort: Lemborexant 10 mg; Day 1: SpO2 is <90%; Test type: Other; p = 0.472, mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.312, 95% CI 2-sided [-0.558 to 1.181]
Statistical Analysis 2: Comparison: OSA Cohort: Placebo vs OSA Cohort: Lemborexant 10 mg; Day 1: SpO2 is <85%; Test type: Other; p = 0.479, mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.067, 95% CI 2-sided [-0.124 to 0.258]
Statistical Analysis 3: Comparison: OSA Cohort: Placebo vs OSA Cohort: Lemborexant 10 mg; Day 1: SpO2 is <80%; Test type: Other; p = 0.852, mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.002, 95% CI 2-sided [-0.019 to 0.023]
Statistical Analysis 4: Comparison: OSA Cohort: Placebo vs OSA Cohort: Lemborexant 10 mg; Day 8: SpO2 is <90%; Test type: Other; p = 0.733, mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.088, 95% CI 2-sided [-0.431 to 0.607]
Statistical Analysis 5: Comparison: OSA Cohort: Placebo vs OSA Cohort: Lemborexant 10 mg; Day 8: When SpO2 is <85%; Test type: Other; p = 0.518, mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LSM difference = 0.056, 95% CI 2-sided [-0.117 to 0.228]
Statistical Analysis 6: Comparison: OSA Cohort: Placebo vs OSA Cohort: Lemborexant 10 mg; Day 8: SpO2 is <80%; Test type: Other; p = 0.576, mixed effect model — P-Value was at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.006, 95% CI 2-sided [-0.015 to 0.026]

9. Secondary Outcome: OSA Cohort: Percentage of Participants With at Least One Incident of SpO2 <90% for at Least 30 Seconds During TST on Day 1 and Day 8 of Treatment
Description: as for outcome 6
Time Frame: Day 1 and Day 8
Population: as for outcome 3
Measure: Number; unit: percentage of participant
Arm/Group | OSA Cohort: Placebo | OSA Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 37 | 37
percentage of participant
  Day 1: SpO2 <90% | 67.6 | 75.7
  Day 8: SpO2 <90% | 75.7 | 83.8

ADVERSE EVENTS:
Time Frame: Baseline up to end of follow up visit (up to 67 days)
Description: Safety analysis set included group of participants who received study drug and had at least 1 postdose safety assessment.
Arm/Group | HV Cohort: Placebo | HV Cohort: Lemborexant 10 mg | HV Cohort: Lemborexant 25 mg | OSA Cohort: Placebo | OSA Cohort: Lemborexant 10 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/17 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/17 | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 1/16 | 1/16 | 4/17 | 5/38 | 6/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HV Cohort: Placebo (N=16) | HV Cohort: Lemborexant 10 mg (N=16) | HV Cohort: Lemborexant 25 mg (N=17) | OSA Cohort: Placebo (N=38) | OSA Cohort: Lemborexant 10 mg (N=38)
Photopsia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT03471871/Prot_002.pdf
  • Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT03471871/SAP_003.pdf